CLINICAL TRIAL: NCT02231450
Title: Interventional, Open-label, Three-group Study to Determine the Pharmacokinetic Properties of Single Oral Dosing of Lu AE58054 in Patients With Hepatic Impairment (Mild and Moderate) and in Healthy Subjects
Brief Title: Pharmacokinetics Properties of Single Oral Dosing of Lu AE58054 in Subjects With Hepatic Impairment (Mild and Moderate) and in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15877A; 2013-004449-18 (EudraCT Number)
Record Dates: First submitted 2014-09-01; First posted 2014-09-04 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Heptic Impairment
Keywords: AE58054; Hepatic impairment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Patients with mild hepatic impairment (Group1) (Experimental): 8 patients with mild hepatic impairment will be administered a single oral dose of 60 mg Lu AE58054
  Interventions: Drug: Lu AE58054 encapsulated film-coated tablets
- Patients with moderate hepatic impairment (Group 2) (Experimental): 8 patients with moderate hepatic impairment will be administered a single oral dose of 60 mg Lu AE58054.
  Interventions: Drug: Lu AE58054 encapsulated film-coated tablets
- Healthy subjects (Group 3) (Experimental): 8 healthy subjects will be administered a single oral dose of 60 mg Lu AE58054.
  Interventions: Drug: Lu AE58054 encapsulated film-coated tablets

INTERVENTIONS:
Drug: Lu AE58054 encapsulated film-coated tablets

SUMMARY:
The purpose of this study is to assess the impact of mild to moderate hepatic impairment on the pharmacokinetics of Lu AE58054 following a single oral dose of Lu AE58054

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 40 and 65 years (inclusive) with a body mass index between 19 and 32 kg/m2 (inclusive).
* Group 1: Patients with mild hepatic impairment (Child-Pugh's Criteria A, score 5-6)
* Group 2: Patients with moderate hepatic impairment (Child-Pugh's Criteria B, score 7-9)
* Group 3: Healthy subjects with normal hepatic function

Other pre-defined inclusion and exclusion criteria may apply.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-07; Primary Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Area under the Lu AE58054 plasma concentration-time curve from time zero to infinity (AUC0-inf) | 0 to 96 hours
Maximum observed plasma concentration (Cmax) of Lu AE58054 | 0 to 96 hours

SECONDARY OUTCOMES:
Absolute values and changes from baseline in safety variables (Adverse events, clinical safety laboratory tests, vital signs, weight, and ECG) | Screening to day 11

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (1):
- APEX GmbH, Munich, Germany